CLINICAL TRIAL: NCT03292952
Title: A Multicenter, Dose-Optimized, Double-Blind, Randomized, Placebo-Controlled, Parallel Efficacy Laboratory Classroom Study With KP415 in Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: KP415 Classroom Study in Children (6-12 Years of Age) With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zevra Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KP415.E01
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-03

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: 3-week, open-label dose-optimization phase followed by a 1-week randomized, double-blind treatment phase
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-blind KP415 (Experimental): KP415 (serdexmethylphenidate [SDX] Cl/ d-methylphenidate [d-MPH] HCl) oral capsule:
  28/6 mg SDX/d-MPH (molar equivalent to 20 mg d-MPH HCl), 42/9 mg SDX/d-MPH (molar equivalent to 30 mg d-MPH HCl), 56/12 mg SDX/d-MPH (molar equivalent to 40 mg d-MPH HCl)
  Interventions: Drug: KP415 oral capsule
- Double-blind Placebo (Placebo Comparator): Placebo oral capsule
  Interventions: Drug: Placebo oral capsule
- Open-Label KP415 (Experimental): KP415 (serdexmethylphenidate [SDX] Cl/ d-methylphenidate [d-MPH] HCl) oral capsule:
  28/6 mg SDX/d-MPH (molar equivalent to 20 mg d-MPH HCl), 42/9 mg SDX/d-MPH (molar equivalent to 30 mg d-MPH HCl), 56/12 mg SDX/d-MPH (molar equivalent to 40 mg d-MPH HCl)
  Interventions: Drug: KP415 oral capsule

INTERVENTIONS:
Drug: KP415 oral capsule — Daily dose
  Arms: Double-blind KP415; Open-Label KP415
Drug: Placebo oral capsule — Daily dose
  Arms: Double-blind Placebo

SUMMARY:
The study is a multicenter, dose-optimized, double-blind, randomized, placebo-controlled, parallel efficacy laboratory classroom study with KP415 in children with Attention-Deficit/Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
The study will consist of a Screening Period, an Open-Label Dose Optimization Phase, a Double-Blind Treatment Phase and a Follow-Up Visit, as follows:

* Screening Period: Subjects will undergo a screening period up to 49 days prior to entering into the Open-Label Dose Optimization Phase.
* Open-Label Dose Optimization Phase: During the Dose Optimization Phase, subjects will be titrated to doses of 20, 30 or 40 mg KP415 based on tolerability and best individual dose-response in the opinion of the Investigator.
* Double-Blind Treatment Phase: Eligible subjects will be randomized to receive single daily doses of KP415 or Placebo for 7 days according to a randomization schedule. The dose of KP415 given in the Treatment Phase will be the same as the optimized dose of KP415 at the end of the Dose Optimization Phase. All subjects will receive their assigned treatment daily for 7 days. The dose will be the same at each day of the Treatment Period. Efficacy and safety assessments will be performed after the last dose of the Treatment Period.
* Follow-Up Visit: 3 ±2 days after administration of the last dose of the Treatment Phase, subjects will enter a Follow-Up Visit to evaluate safety parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD (combined, inattentive, or hyperactive/impulsive presentation) per clinical evaluation and confirmed by the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
2. Subject must have a score of at least 3 (mildly ill) on the clinician-administered Clinical Global Impressions-Severity (CGI-S) scale.
3. Subject, subject's parent/legal guardian and caregiver (if applicable) must understand and be willing and able to comply with all study procedures and visit schedule.

Exclusion Criteria:

1. Subject with any clinically significant chronic medical condition that may interfere with the participant's ability to participate in the study.
2. Subject has any diagnosis of bipolar I or II disorder, major depressive disorder, conduct disorder, obsessive-compulsive disorder, any history of psychosis, autism spectrum disorder, disruptive mood dysregulation disorder (DMDD), intellectual disability, Tourette's Syndrome, confirmed genetic disorder with cognitive and/or behavioral disturbances.
3. Subject has evidence of any chronic disease of the central nervous system (CNS) such as tumors, inflammation, seizure disorder, vascular disorder, potential CNS related disorders that might occur in childhood, or history of persistent neurological symptoms attributable to serious head injury.
4. Subject has a current (last month) psychiatric diagnosis other than specific phobia, motor skills disorders, oppositional defiant disorder, sleep disorders, elimination disorders, adjustment disorders, learning disorders, or communication disorders. Participants with school phobia or separation anxiety will not be eligible.
5. Subject has any history of attempted suicide or clinically significant suicidal ideation or subject has a C-SSRS score for suicidal ideation ≥2.
6. Subject has any clinically significant unstable medical abnormality, chronic disease, or a history of a clinically significant abnormality of the cardiovascular, gastrointestinal, respiratory, hepatic, or renal systems, or a disorder or history of a condition that may interfere with drug absorption, distribution, metabolism, or excretion of study drug.
7. Subject has a history or presence of abnormal ECGs.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott H Kollins, PhD, Principal Investigator — Duke Clinical Research Institute
Locations (5):
- United States (5):
  - Meridien Research, Bradenton, Florida
  - Meridien Research, Maitland, Florida
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Duke University Medical Center, Durham, North Carolina
  - Bayou City Research, Ltd., Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label KP415: Open-label titration with KP415 capsule 20, 30, or 40 mg once-daily for 3 weeks
- Double-Blind KP415: KP415 oral capsule 20, 30 or 40 mg
  KP415 oral capsule: Daily dose
Period: Open-Label Dose Optimization
Arm/Group | Open-Label KP415 | Double-Blind KP415 | Double-Blind Placebo
Started | 155 | 0 (All subjects were treated with open-label KP415 during the Open-Label Phase) | 0 (All subjects were treated with open-label KP415 during the Open-Label Phase)
Completed | 150 | 0 | 0
Not Completed | 5 | 0 | 0
Period: Double-Blind Treatment Phase
Arm/Group | Open-Label KP415 | Double-Blind KP415 | Double-Blind Placebo
Started | 0 (Subjects were randomized to the double-blind Treatment Phase after Open-Label Dose Optimization) | 74 | 76
Completed | 0 | 74 | 75
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment: KP415 oral capsule 20, 30 or 40 mg
  KP415 oral capsule: Daily dose
- Placebo Treatment: Placebo oral capsule
  Placebo oral capsule: Daily dose
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.6 (1.6) | 9.6 (1.5) | 9.6 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 44 | 48 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 20 | 40
  Not Hispanic or Latino | 54 | 56 | 110
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 31 | 56
  White | 38 | 38 | 76
  More than one race | 6 | 4 | 10
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 74 | 76 | 150

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) Combined Scores
Description: The SKAMP scale is a validated rating of subjective impairment of classroom behaviors in children with ADHD. It comprises 13 items (grouped under the subcategories of attention, deportment, quality of work, and compliance) on which subjects are rated according to a 7-point scale (0 = normal to 6 = maximal impairment) by trained study personnel (Swanson 1998). The SKAMP-C score was obtained by summing the rating values for each of the 13 items (range: 0-78), with higher scores indicating greater impairment.
Time Frame: Average of all time points during the full laboratory classroom day, which occurred on Day 7 (Day 28 of the overall study) of the Treatment Phase
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 74 | 75
score on a scale | -4.87 (0.62) | 0.536 (0.70)
Statistical Analysis 1: Comparison: Active Treatment vs Placebo Treatment; Test type: Superiority; p < 0.001, ANCOVA

2. Secondary Outcome: Change From Baseline in Permanent Product Measure of Performance (PERMP) Rating Scale, Number of Problems Attempted (PERMP-A)
Description: The PERMP is an adjusted math test designed to assess attention in children with ADHD (Swanson 1999). The test measures attention through a subject's ability to initiate, self-monitor, and complete the math test. A Placement PERMP was performed early in the trial to assure that subjects could complete at least the basic level of math problems and to determine the appropriate level of math to be assigned during the remainder of the study. The PERMP is an individually calibrated 5-page mathematics worksheet consisting of 400 problems. PERMP-A scores document the number of problems attempted, from 0 to 400, and thus higher scores represent a better outcome.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind KP415 | Double-Blind Placebo
Number analyzed (Participants) | 74 | 75
score on a scale | 25.82 (3.44) | 2.25 (3.05)

ADVERSE EVENTS:
Time Frame: 5 weeks
Groups:
- Open-Label KP415: 3-week titration period to identify an optimal dose of KP415 (serdexmethylphenidate [SDX] Cl/ d-methylphenidate [d-MPH] HCl) oral capsule, once-daily:
  28/6 mg SDX/d-MPH (molar equivalent to 20 mg d-MPH HCl), 42/9 mg SDX/d-MPH (molar equivalent to 30 mg d-MPH HCl), 56/12 mg SDX/d-MPH (molar equivalent to 40 mg d-MPH HCl)
- Double-Blind KP415: Optimized dose of KP415 (serdexmethylphenidate [SDX] Cl/ d-methylphenidate [d-MPH] HCl) oral capsule, once-daily:
  28/6 mg SDX/d-MPH (molar equivalent to 20 mg d-MPH HCl), 42/9 mg SDX/d-MPH (molar equivalent to 30 mg d-MPH HCl), 56/12 mg SDX/d-MPH (molar equivalent to 40 mg d-MPH HCl)
- Double-Blind Placebo: Double-Blind Placebo, once-daily
Arm/Group | Open-Label KP415 | Double-Blind KP415 | Double-Blind Placebo
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/74 | 0/76
Other Adverse Events (participants affected / at risk) | 104/155 | 13/74 | 6/76
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label KP415 (N=155) | Double-Blind KP415 (N=74) | Double-Blind Placebo (N=76)
Headache (Nervous system disorders) | 12 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 15 | 3 | 1
Insomnia (Psychiatric disorders) | 24 | 2 | 1
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Affect lability (Psychiatric disorders) | 18 | 1 | 1
Irritability (Psychiatric disorders) | 12 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 38 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 1 | 1
Dizziness (Nervous system disorders) | 4 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 2 | 4
Fatigue (Gastrointestinal disorders) | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT03292952/Prot_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT03292952/SAP_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Addendum (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT03292952/SAP_003.pdf